CLINICAL TRIAL: NCT02758184
Title: Effectiveness of ROTEM-based Coagulation Surveillance on Reducing Blood Product Utilization During Complex Spine Surgery: A Prospective Randomized Study
Brief Title: Effectiveness of ROTEM-based Coagulation Surveillance on Reducing Blood Product Utilization During Complex Spine Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00070817
Record Dates: First submitted 2016-04-19; First posted 2016-05-02 (Estimated); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-03

CONDITIONS: Spine Surgery; Rotational Thrombo-elastometry (ROTEM)

ARMS (2):
- ROTEM Group (Experimental): Patients who are randomized to receive ROTEM
  Interventions: Device: ROTEM-based coagulation monitoring; Procedure: Spine surgery
- Control Group (Other): Patients who are randomized not to receive ROTEM
  Interventions: Procedure: Spine surgery

INTERVENTIONS:
Device: ROTEM-based coagulation monitoring
  Arms: ROTEM Group
Procedure: Spine surgery

SUMMARY:
The Purpose of this study is to identify added value of Rotational thrombo-elastometry (ROTEM) intra-operative coagulation surveillance on reducing blood product use during major reconstructive spine surgery.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effectiveness of intra-operative ROTEM-based coagulation monitoring on reducing total blood product use during complex spine surgery.

The primary outcome will include estimated blood losses and blood product utilization during and after surgery (48 hours).

Secondary outcomes also include hospital length of stay, and cost analysis of the 2 methodologies.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 80 years old.
2. Elective spine surgery cases, with a traditional open posterior approach and involving fusion of at least 5 levels.
3. Normal coagulation profile (PT/INR, aPTT) and normal platelets count on pre-operative evaluation.
4. Preoperative hemoglobin Level >10 g/dl.
5. OR time > 4 hours.
6. No contraindication for the use of anti-fibrinolytic therapy (Tranexamic acid).

Exclusion Criteria:

1. Age < 18 or age > 80 years old.
2. Anterior spine surgeries or posterior spine surgeries involving <5 levels.
3. Minimally invasive spine surgeries.
4. Patients with known coagulopathies or bleeding tendencies or patients with abnormal coagulation laboratory values at baseline.
5. Patients with Hemoglobin level of <10 g/dl on preoperative baseline laboratory values.
6. Trauma and Emergency spine surgeries.
7. Patients with spine malignancy diagnosis, either primary or metastatic.
8. OR time < 4 hours.
9. Patients who refuse to use allogenic blood products.
10. Patients with contraindications for the use of anti-fibrinolytic therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Mendoza-Lattes, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Rotational Thrombo-elastometry (ROTEM) Group: Patients who are randomized to receive ROTEM
  ROTEM-based coagulation monitoring
  Spine surgery
- Control Group: Patients who are randomized not to receive ROTEM
  Spine surgery
Period: Overall Study
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (14.0) | 61.2 (7.8) | 60.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 7 | 7 | 14
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Estimated Blood Loss (mL)
Time Frame: during surgery (up to approximately 10 hours)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 11 | 10
mL | 2318.8 (1629.3) | 3350.0 (1494.6)
Statistical Analysis 1: Comparison: Rotational Thrombo-elastometry (ROTEM) Group vs Control Group; Test type: Other; p = 0.15, ANOVA; Mean Difference (Final Values) = 1031.2, Standard Error of Mean 681.7

2. Primary Outcome: Total Number of Units of Packed Red Blood Cells (PRBCs) Transfused
Time Frame: up to 48 hours after surgery
Measure: Mean (Standard Deviation); unit: units of PRBCs
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 11 | 10
units of PRBCs | 2.81 (1.99) | 5.00 (3.59)

3. Secondary Outcome: Length of Hospital Stay After Surgery
Time Frame: typically 5-7 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 11 | 10
days | 6.3 (1.4) | 6.2 (3.1)

4. Secondary Outcome: Cost Analysis, as Measured by Total Dollar Value of Blood Products Used
Time Frame: during surgery (up to approximately 10 hours)
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 11 | 10
US dollars | 1123.00 (1078.60) | 1998.70 (2020.70)

5. Secondary Outcome: Amount of Recovered Blood Transfused During the Procedure (mL)
Time Frame: during surgery (up to approximately 10 hours)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 11 | 10
mL | 476.3 (434.3) | 879.4 (755.1)

6. Secondary Outcome: Drain Output (mL)
Time Frame: first 24 hours after surgery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 11 | 10
mL | 587.5 (362.7) | 757.8 (335.3)

7. Secondary Outcome: Amount of Blood Products Transfused, Measured in Units
Time Frame: during surgery (up to approximately 10 hours)
Measure: Mean (Standard Deviation); unit: units of blood product
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 11 | 10
units of blood product | 4.81 (4.68) | 7.80 (8.30)

8. Secondary Outcome: Amount of Blood Products Transfused, Measured in Units
Time Frame: 48 hours following surgery
Measure: Mean (Standard Deviation); unit: units of blood product
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 11 | 10
units of blood product | 0.54 (0.93) | 1.20 (1.39)

9. Secondary Outcome: Change in Hemoglobin (g/dL)
Description: Reporting the change in hemoglobin from baseline to approximately 10 hours.
Time Frame: Baseline and approximately every 2 hours during surgery (up to approximately 10 hours)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 11 | 10
g/dL | -2.56 (1.74) | -2.78 (1.02)

10. Secondary Outcome: Change in Platelet Count
Description: Reporting the change in platelet count from baseline to approximately 10 hours.
Time Frame: Baseline and approximately every 2 hours during surgery (up to approximately 10 hours)
Measure: Mean (Standard Deviation); unit: platelets/uL
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 11 | 10
platelets/uL | -74.0 (66.6) | -57.1 (34.2)

11. Secondary Outcome: Change in Prothrombin Time
Time Frame: Baseline and approximately every 2 hours during surgery (up to approximately 10 hours)
Population: Data not collected.
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in International Normalized Ratio (PT/INR)
Time Frame: Baseline and approximately every 2 hours during surgery (up to approximately 10 hours)
Population: Data not collected.
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in Activated Partial Thromboplastin Time (aPTT)
Time Frame: Baseline and approximately every 2 hours during surgery (up to approximately 10 hours)
Population: Data not collected.
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Fibrinogen (g/L)
Time Frame: Baseline and approximately every 2 hours during surgery (up to approximately 10 hours)
Population: Data not collected.
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 48 hours after surgery.
Description: Only Adverse Events related to the study are reported.
Arm/Group | Rotational Thrombo-elastometry (ROTEM) Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT02758184/Prot_SAP_000.pdf